CLINICAL TRIAL: NCT06036472
Title: Impact of Periodontal Therapy on Mental Health Parameters in Patients With Major Depression and Periodontitis: a Pilot Randomized Controlled Clinical Trial.
Brief Title: Impact of Periodontal Therapy on Mental Health Parameters
Acronym: LeakBrainRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URI 107-260623
Record Dates: First submitted 2023-07-26; First posted 2023-09-14 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis; Depression
MeSH Terms: conditions — Periodontitis; Depression | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subgingival therapy (Experimental): Participant will receive standard periodontal treatment consisting of two sessions of supra- and subgingival debridement (steps 1 and 2) under local anesthesia following current guidelines for periodontal therapy in patients with periodontitis (Herrera et al., 2022; Sanz et al., 2020). The use of chlorhexidine (0.12%) and cetylpyridinium chloride (0.05%) mouthwash will be prescribed twice a day for 15 days (Perio-Aid®, Dentaid, Barcelona, Spain). If needed, hopeless teeth might be extracted during this step.
  Interventions: Procedure: Standard periodontal therapy (steps 1 & 2)
- Supragingival therapy (Other): Periodontal treatment consisting of two sessions of supragingival debridement with anesthesia (step 1) and administration of a placebo mouthwash (FluorAid®, Dentaid, Barcelona, Spain), twice a day for 15 days.
  Interventions: Procedure: supragingival debridement with anesthesia (step 1)

INTERVENTIONS:
Procedure: Standard periodontal therapy (steps 1 & 2) — participant will receive standard periodontal treatment consisting of two sessions of supra- and subgingival debridement (steps 1 and 2) under local anesthesia following current guidelines for periodontal therapy in patients with periodontitis (Herrera et al., 2022; Sanz et al., 2020). The use of chlorhexidine (0.12%) and cetylpyridinium chloride (0.05%) mouthwash will be prescribed twice a day for 15 days (Perio-Aid®, Dentaid, Barcelona, Spain). If needed, hopeless teeth might be extracted during this step.
  Arms: Subgingival therapy
Procedure: supragingival debridement with anesthesia (step 1) — periodontal treatment consisting of two sessions of supragingival debridement with anesthesia (step 1) and administration of a placebo mouthwash (FluorAid®, Dentaid, Barcelona, Spain), twice a day for 15 days.
  Arms: Supragingival therapy

SUMMARY:
Objectives: Primary: To determine the efficacy of periodontal treatment on mental health outcomes in patients with major depression and periodontitis. Secondary: To identify the effect of periodontal treatment on oral, periodontal, and fecal metagenomic microbiomes, and on systemic levels of inflammation (bacterial, viral, and fungal) and their impact on mental health outcomes.

Material and method:

A 6-month pilot randomized controlled clinical trial is designed. The study will be conducted in patients with moderate or severe DM (Patient Health Questionnaire-9 [PHQ-9] index of 9 or higher) and stage III-IV periodontitis who will be assigned to two different interventions:

* Test group: standard periodontal treatment consisting of two sessions of supragingival and subgingival debridement (steps 1 and 2) under local anesthesia.
* Control group: periodontal treatment consisting of two sessions of supragingival debridement (step 1) under local anesthesia.

The study will consist of 6 visits:

* Screening visit (v0)
* Baseline visit (v1):

  * In the mental health center: patients will receive a structured clinical interview for the DSM-IV (SCID) and the patient will fill out a series of specific scales on a study-specific electronic device [Beck Depression Inventory (BDI); UCLA Loneliness Scale, Center for Epidemiologic Studies Depression scale [CES-D]; Childhood Trauma Questionnaire short form (CTQ-SF); The World Health Organization Quality of Life questionnaire (WHOQOL); Hamilton scale (HAM-D17); Global Assessment of Functioning (GAF) Scale].
  * At the UCM School of Dentistry: patients will receive a complete periodontal examination (clinical and radiographic). A subgingival microbiological sample, a saliva sample and a blood sample will also be taken.
  * At the participant's home: the stool samples will be deposited by the participants at home in the specific collection vial.
* Intervention visits (v2-3): Two periodontal treatment sessions (test or control) will be carried out one week apart.
* Re-evaluation visit (v4): Six weeks after treatment, all periodontal clinical variables will be recorded.
* Follow-up visits at 3 and 6 months: after periodontal treatment, all the variables recorded at the baseline visit will be taken

Statistical analysis:

Periodontal treatment (test/control) will be considered as the independent variable and the Hamilton scale (HAM-D17) will be considered the primary response variable. The rest of the variables will be considered as secondary variables. A crude bivariate analysis of comparison of means or proportions will be carried out depending on the nature of the variable. In addition, crude and adjusted regression models will be performed.

ELIGIBILITY:
5.3.1. Inclusion criteria:

* Age greater or equal to 18 years.
* Patients with moderate or severe major depression, without severe suicide ideation, as characterized by the Patient Health Questionnaire (PHQ)-9 index (values of 9 or greater) and by the Structured Clinical Interview for DSM-5 - (SCID) will be selected.
* Subjects with periodontitis stages III or IV, according to the 2018 Classification on periodontal and peri-implant diseases (Papapanou et al., 2018).

5.3.2. Exclusion criteria:

* Pregnant or breastfeeding women.
* Diabetes mellitus.
* Chronic conditions: HIV infection, chronic intake of NSAIDs.
* Comorbidity with other mental disorders: eating disorders, borderline personality disorders, bipolar disorders, schizophrenia and related disorders, and/or any mental serious disease other than major depression.
* Severe suicide ideation.
* Smokers of 10 or more cigarettes per day.
* Patients who had received periodontal treatment for periodontitis in the last year.
* Presence of necrotizing periodontal diseases.
* Presence of less than 3 teeth per quadrant.
* Antibiotic use in the last 6 months prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton scale (HAM-D17) | Baseline
  Range: 0 to 52. The higher the score, the more severethe depressive symptoms
Hamilton scale (HAM-D17) | 3 months
  Range: 0 to 52. The higher the score, the more severethe depressive symptoms
Hamilton scale (HAM-D17) | 6 months
  Range: 0 to 52. The higher the score, the more severethe depressive symptoms

SECONDARY OUTCOMES:
Childhood Trauma Questionnaire short form (CTQ-SF) | Baseline
  Range: 25 to 125. A higherscore means more (and worst) traumatic experience
Childhood Trauma Questionnaire short form (CTQ-SF) | 3 months
  Range: 25 to 125. A higherscore means more (and worst) traumatic experience
Childhood Trauma Questionnaire short form (CTQ-SF) | 6 months
  Range: 25 to 125. A higherscore means more (and worst) traumatic experience
UCLA Loneliness Scale (Spanish version) | Baseline
  Range: 20 to 80. Higher scores indicatehigher levels of loneliness
UCLA Loneliness Scale (Spanish version) | 3 months
  Range: 20 to 80. Higher scores indicatehigher levels of loneliness
UCLA Loneliness Scale (Spanish version) | 6 months
  Range: 20 to 80. Higher scores indicatehigher levels of loneliness
The World Health Organization Quality of Life questionnaire (WHOQOL) | Baseline
  Range: o to100. A higher score means better quality of life.
The World Health Organization Quality of Life questionnaire (WHOQOL) | 3 months
  Range: o to100. A higher score means better quality of life.
The World Health Organization Quality of Life questionnaire (WHOQOL) | 6 months
  Range: o to100. A higher score means better quality of life.
Beck Depression Inventory (BDI) | Baseline
  Range: 0 to 63. A higher score means more severe-depressive symptomatology
Beck Depression Inventory (BDI) | 3 months
  Range: 0 to 63. A higher score means more severe-depressive symptomatology
Beck Depression Inventory (BDI) | 6 months
  Range: 0 to 63. A higher score means more severe-depressive symptomatology
Centre for Epidemiologic Studies Depression scale [CES-D] | Baseline
  Range: 0 to 60. Higher scores indicate the presence of more severe symptomatology
Centre for Epidemiologic Studies Depression scale [CES-D] | 3 months
  Range: 0 to 60. Higher scores indicate the presence of more severe symptomatology
Centre for Epidemiologic Studies Depression scale [CES-D] | 6 months
  Range: 0 to 60. Higher scores indicate the presence of more severe symptomatology
Global Assessment of Functioning (GAF) Scale | Baseline
  Range: 1 to 100. A higher scoremeans better functioning. A score of 0 means Inadequate information.
Global Assessment of Functioning (GAF) Scale | 3 months
  Range: 1 to 100. A higher scoremeans better functioning. A score of 0 means Inadequate information.
Global Assessment of Functioning (GAF) Scale | 6 months
  Range: 1 to 100. A higher scoremeans better functioning. A score of 0 means Inadequate information.

OTHER OUTCOMES:
Plaque index | Baseline
  presence/absence
Plaque index | 3 months
  presence/absence
Plaque index | 6 months
  presence/absence
Bleeding on probing | Baseline
  Assessed dichotomously within 15 seconds after probing
Bleeding on probing | 3 months
  Assessed dichotomously within 15 seconds after probing
Bleeding on probing | 6 months
  Assessed dichotomously within 15 seconds after probing
Suppuration on probing | Baseline
  Assessed dichotomously post-probing
Suppuration on probing | 3 months
  Assessed dichotomously post-probing
Suppuration on probing | 6 months
  Assessed dichotomously post-probing
Probing depth | Baseline
  Defined as the distance in mm between the bottom of the pocket and the gingival margin
Probing depth | 3 months
  Defined as the distance in mm between the bottom of the pocket and the gingival margin
Probing depth | 6 months
  Defined as the distance in mm between the bottom of the pocket and the gingival margin
Recession | Baseline
  defined as the distance in mm between the amelocemental boundary and the gingival margin.
Recession | 3 months
  defined as the distance in mm between the amelocemental boundary and the gingival margin.
Recession | 6 months
  defined as the distance in mm between the amelocemental boundary and the gingival margin.
Number of teeth lost | Baseline
Number of teeth lost | 3 months
Number of teeth lost | 6 months
Microbiological outcomes | Baseline
  Subgingival biofilm samples will be taken from samples of gingival crevicular fluid. DNA samples will be frozen at -20°C and preserved until further analysis by quantitative polymerase chain reaction (q-PCR) and 16S rRNA sequencing, using the Illumina MiSeq platform
Microbiological outcomes | 3 months
  Subgingival biofilm samples will be taken from samples of gingival crevicular fluid. DNA samples will be frozen at -20°C and preserved until further analysis by quantitative polymerase chain reaction (q-PCR) (Marín et al., 2019) and 16S rRNA sequencing, using the Illumina MiSeq platform
Microbiological outcomes | 6 months
  Subgingival biofilm samples will be taken from samples of gingival crevicular fluid. DNA samples will be frozen at -20°C and preserved until further analysis by quantitative polymerase chain reaction (q-PCR) (Marín et al., 2019) and 16S rRNA sequencing, using the Illumina MiSeq platform
Plasma levels of inflammatory mediators | Baseline
  Interleukin-1β, Tumor Necrosis Factor-α, prostaglandin-E2, C reactive protein, D-Lactate and intestinal-type fatty acid binding protein 2 [FABP2]), lipopolysaccharide (LPS). matrix metalloproteinase (MMP)-9 levels, S-100B protein levels, quinolinic acid levels, and the ratio between kynurenic and quinolinic acid
Plasma levels of inflammatory mediators | 3 months
  Interleukin-1β, Tumor Necrosis Factor-α, prostaglandin-E2, C reactive protein, D-Lactate and intestinal-type fatty acid binding protein 2 [FABP2]), lipopolysaccharide (LPS). matrix metalloproteinase (MMP)-9 levels, S-100B protein levels, quinolinic acid levels, and the ratio between kynurenic and quinolinic acid
Plasma levels of inflammatory mediators | 6 months
  Interleukin-1β, Tumor Necrosis Factor-α, prostaglandin-E2, C reactive protein, D-Lactate and intestinal-type fatty acid binding protein 2 [FABP2]), lipopolysaccharide (LPS). matrix metalloproteinase (MMP)-9 levels, S-100B protein levels, quinolinic acid levels, and the ratio between kynurenic and quinolinic acid
Saliva samples | Baseline
  Oral microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences will be compared to phylogenetic and functional databases to obtain taxonomic and functional profiles.
Saliva samples | 3 months
  Oral microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences will be compared to phylogenetic and functional databases to obtain taxonomic and functional profiles.
Saliva samples | 6 months
  Oral microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences will be compared to phylogenetic and functional databases to obtain taxonomic and functional profiles.
Stool samples | Baseline
  Gut microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences will be compared to phylogenetic and functional databases to obtain taxonomic and functional profiles.
Stool samples | 3 months
  Gut microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences will be compared to phylogenetic and functional databases to obtain taxonomic and functional profiles.
Stool samples | 6 months
  Gut microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences will be compared to phylogenetic and functional databases to obtain taxonomic and functional profiles.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Dentistry, University Complutense of Madrid (UCM), Madrid
  - Instituto de Psiquiatría y Salud Mental, Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: Undecided